CLINICAL TRIAL: NCT05870839
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of VXCO-100 in Healthy Adults in the United States
Brief Title: Study of VXCO-100, a SARS-CoV Candidate Vaccine in Healthy Adults in the United States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaccine Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VC 101
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: SARS-CoV; SARS-CoV-2
Keywords: Covid-19; SARS-CoV-2; Coronavirus; Vaccine; Sarbecoviruses; Covid
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- VXCO-100 Group 1 (Experimental): Participants 18-55 years of age will receive VXCO-100 at Dose Level 1 via intramuscular (IM) injection
  Interventions: Biological: VXCO-100
- VXCO-100 Group 2 (Experimental): Participants 18-55 years of age will receive VXCO-100 at Dose Level 2 via intramuscular (IM) injection
  Interventions: Biological: VXCO-100
- VXCO-100 Group 3 (Experimental): Participants 18-55 years of age will receive VXCO-100 at Dose Level 3 via intramuscular (IM) injection
  Interventions: Biological: VXCO-100
- VXCO-100 Group 4 (Experimental): Participants 56+ years of age will receive VXCO-100 at Dose Level 1 via intramuscular (IM) injection
  Interventions: Biological: VXCO-100
- VXCO-100 Group 5 (Experimental): Participants 56+ years of age will receive VXCO-100 at Dose Level 2 via intramuscular (IM) injection
  Interventions: Biological: VXCO-100
- VXCO-100 Group 6 (Experimental): Participants 56+ years of age will receive VXCO-100 at Dose Level 3 via intramuscular (IM) injection
  Interventions: Biological: VXCO-100

INTERVENTIONS:
Biological: VXCO-100 — Sterile liquid for injection

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of ascending dose levels of VXCO-100 in healthy adults.

DETAILED DESCRIPTION:
This is a phase 1, multisite clinical trial to evaluate the safety and immunogenicity of 3 dose levels of VXCO-100 in healthy adult volunteers.

Participants will be vaccinated with 1 dose of VXCO-100 on Day 1. A subset of participants will be offered an optional interim boost at month 3.

Safety will be evaluated 1) before proceeding to a higher dose level and 2) prior to enrollment of participants aged 56 years and older at a particular dose level.

ELIGIBILITY:
Inclusion Criteria

A participant must meet all the following criteria to be eligible for the study:

* Adults ages 18 years and older.
* Judged by the investigator to be healthy based on participant-reported medical history, physical examination, vital signs, and laboratory assessment.
* Able to provide written informed consent.
* Willing to disclose prior COVID-19 vaccination status.
* Willing to disclose prior participant-reported SARS-CoV-2 infection status.
* Prior receipt of at least 3 injections with a COVID-19 mRNA vaccine with the most recent dose at least 6 months prior to enrollment.
* Willing to comply with all study procedures during the follow-up period of approximately 12 or 24 months, depending on number of doses received.
* Body mass index of ≤ 40 kg/m2 within 30 days prior to enrollment
* Electrocardiogram (ECG) without clinically significant abnormalities. Laboratory Criteria within 30 days before enrollment
* White blood cells (WBC) and differential within institutional normal range or accompanied by the site Principal Investigator (PI) or designee approval.
* Total lymphocyte count ≥ 800 cells/µL.
* Platelets between 125,000 and 500,000 cells/µL.
* Hemoglobin within institutional normal range or accompanied by the PI or designee approval.
* Alanine aminotransferase (ALT) ≤ 1.25 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) ≤ 1.25 x institutional ULN.
* Serum creatinine ≤ 1.1 x institutional ULN.
* Ferritin, iron and TIBC within institutional normal range or accompanied by the PI or designee approval.

For participants of childbearing potential:

* Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on the day of enrollment.
* Must agree to avoid pregnancy from 21 days prior to study Day 1 until at least 90 days after last study vaccination.

Exclusion Criteria

A participant will be excluded if one or more of the following conditions apply:

* Known SARS-CoV-2 infection or positive test result within 6 months prior to Day 1.
* Ongoing prophylactic COVID-19 treatment, or monoclonal antibody infusion within 6 months prior to Day 1.
* Any COVID-19 vaccination within 6 months prior to Day 1.
* Exhibits symptoms consistent with COVID-19 as assessed by study clinician such as: fever, dry cough, fatigue, nasal obstruction, runny nose, sore throat, myalgia, diarrhea, shortness of breath or dyspnea within 14 days prior to in Day 1.
* Known close contact (as defined by CDC, 2021a) with someone who has COVID-19 within 14 days prior to Day 1.
* History or presence of self-reported or medically documented significant medical or psychiatric condition(s) as assessed by study clinician, including:
* At high risk of severe COVID-19 disease, such as significant history of COPD or chronic lung disease, chronic kidney disease, serious heart conditions (such as heart failure, coronary artery disease or cardiomyopathies), sickle cell disease, diabetes.
* Clinically significant central nervous system disease such as epilepsy, encephalopathy, or a history of severe mental illness.
* Severe liver and/or kidney diseases, uncontrolled hypertension, or ongoing or highly likely to recur malignancies.
* Ongoing or recent clinically significant history of alcohol or drug abuse.
* Current participation in an interventional clinical study with an investigational drug/biologic/device agent or receipt of any investigational agent within 30 days prior to Day 1.
* Evidence of infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
* History of myocarditis or pericarditis.
* Diagnosed with congenital or acquired immune deficiency, ongoing lymphoma, leukemia, or other clinically significant immune compromising or autoimmune conditions.
* History of known coagulation dysfunction (e.g., coagulation factor deficiency, known thrombocytopenia, platelet dysfunction, coagulation disease, etc.).
* Receipt of any live attenuated vaccine within 30 days, or with any other (non-live) vaccine within 14 days prior to Day 1.
* Received more than 10 days of any systemic immunosuppressants or cytotoxic medications within 30 days prior to Day 1, any within 14 days prior to Day 1 or is anticipating the need for immunosuppressants at any time during participation in the study.
* Received any blood products within 3 months prior to Day 1.
* Donated > 450 mL of whole blood within 30 days prior to Day 1.
* History of unexplained or recurrent anaphylaxis or angioedema, or a history of severe allergic reaction (e.g., anaphylaxis) after a previous dose of any vaccine, or to any component of the study vaccine.
* For participants of childbearing potential: breastfeeding or planning to become pregnant during trial duration.
* Any condition that, in the opinion of the investigator, would (a) pose a health risk to the participant if enrolled or (b) could interfere with evaluation of the study vaccine or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with solicited local adverse events | For 7 days after each product administration
Number and percentage of participants with solicited systemic adverse events | For 7 days after each product administration
Number and percentage of participants with unsolicited and safety laboratory-based adverse events | For 28 days after each product administration
Numbers and percentages of participants with serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs), medically attended adverse events (MAAEs), and adverse events of special interest (AESIs) | For up to 304 days after each product administration

SECONDARY OUTCOMES:
Response rate measured by geometric mean titer of the serum neutralizing antibody (Nab) against the ancestral (Wuhan) strain | At baseline and 21 days after each product administration
Response rate measured by GMT of Nab against selected variants of concern | At baseline and 21 days after each product administration
Numbers and percentages of participants with positive Th1 or Th2 cytokine responses for CD4 and CD8 as measured by multi-parameter intracellular cytokine staining | At baseline and 7 days after each product administration

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ortiz, MD, MS, Principal Investigator — University of Maryland; Nadine Rouphael, MD, Principal Investigator — Emory University; Angela Branche, MD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York

IPD SHARING:
Plan to Share IPD: No